CLINICAL TRIAL: NCT03132688
Title: A Retrospective Study on Safety and Efficacy of Propofol in Small Children
Brief Title: A Study on Safety and Efficacy of Propofol in Small Children Under 2 Years of Age
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Other Study IDs: H1612-136-821
Record Dates: First submitted 2017-02-21; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Heart Rate Low; Anesthesia; Functional
MeSH Terms: conditions — Bradycardia | interventions — Propofol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children < 2 years old: Children under 2 years of age who received intravenous propofol during general anesthesia.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Intravenous administration with dose of 100-200mcg/kg/min

SUMMARY:
This retrospective study the safety and efficacy of intravenous propofol used in children under 2 years of age during general anesthesia for surgery.

DETAILED DESCRIPTION:
EMR review of intravenous propofol used in target controlled infusion method in children under 2 years old.

ELIGIBILITY:
Inclusion Criteria:

* Children under 2 years of age
* Children who received intravenous propofol for maintenance of anesthesia

Exclusion Criteria:

* Children who underwent general anesthesia with inhalational anesthetics

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who underwent surgery From September 2013 to December 2016 , and received intravenous propofol for general anesthesia will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-04-22 (Actual); Study Completion 2017-04-22 (Actual)

PRIMARY OUTCOMES:
Safety: blood pressure | Intraoperative 1 day
  blood pressure
Safety: blood pressure | Intraoperative 7th days
  blood pressure

SECONDARY OUTCOMES:
Bispectral index | Intraoperative
  optimal surgical condition

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided